CLINICAL TRIAL: NCT04806347
Title: TCRαβ+ and CD19+ Depleted Hematopoietic Stem Cell Transplant From Closely Matched Unrelated Donors or Haploidentical Related Donors for Hematologic Diseases in Children and Young Adults
Brief Title: Alpha/Beta T-cell Depleted Blood-forming Stem Cell Transplant From Related or Unrelated Donors for Blood Diseases in Children and Young Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1251; 2020-1251 (Other: HS IRB UW Madison); A536755 (Other: UW Madison); Protocol Version 4 (Other: HS-IRB UW Madison); NCI-2021-02128 (Registry Identifier: NCI CTRP); UW19113 (Other: OnCore ID)
Record Dates: First submitted 2021-03-02; First posted 2021-03-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-07

CONDITIONS: Blood Disease
MeSH Terms: conditions — Hematologic Diseases | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment arm (Experimental): Participants will undergo a conditioning regimen, specific for the original disease, After that peripheral blood stem cell transplant from a haploidentical donor or closely matched unrelated donor, depleted of TCRαβ+ and CD19+ cells using the CliniMACS TCR α/β-biotin and CD19 Systems will be administered intravenously on Day 0 to all participants.
  Interventions: Biological: TCRαβ+/CD19+ depleted Hematopoietic stem cell (HSC) graft; Device: CliniMACS® System

INTERVENTIONS:
Biological: TCRαβ+/CD19+ depleted Hematopoietic stem cell (HSC) graft — After undergoing a disease specific conditioning regimen (standard of care), participants will receive peripheral blood stem cell transplant from a haploidentical donor or closely matched unrelated donor, depleted of TCR αβ+ and CD19+ cells using the CliniMACS TCR α/β-biotin and CD19 Systems.
Device: CliniMACS® System — The CliniMACS Cell Selection System is based on magnetic-activated cell sorting mechanism. The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures.

SUMMARY:
This single institution, phase I clinical trial will determine the safety and feasibility of employing T-cell receptor (TCR) αβ+ and CD19+ (Cluster of Differentiation ) depleted hematopoietic stem cell transplantation (HSCT) using peripheral blood stem cells (PBMC) from closely matched unrelated donors or haploidentical donors to treat non-malignant hematologic diseases in children and young adults. Allogeneic hematopoietic stem cell transplantation has become a curative option for children and adolescents with a variety of otherwise fatal conditions. To reduce the incidence and severity of graft-versus-host disease (GVHD) associated with allogeneic hematopoietic stem cell transplantation, donor grafts are depleted of T cells, either using CD34+ selection or CD3+/CD19+ depletion of grafts. However, these selection processes also deplete the graft of protective cell subsets, such as γδ T cells, natural killer(NK) cells, monocytes and dendritic cells, which play important roles in the immune response to infectious agents. Moreover, the presence of NK cells and γδ T in donor grafts is associated with more rapid immune reconstitution after HSCT transplantation. In order to retain these protective immune cell subsets, this trial will use a novel, highly selective graft engineering process using the Miltenyi CliniMACS system that selectively depletes αβ-T cells and B cells which are responsible for GVHD and Epstein Barr Virus (EBV)-related post-transplantation lymphoproliferative disorder, respectively. Prior to transplantation, patients will be treated with a conditioning regimen, specific for the original disorder. The primary objective of this study is evaluation of the safety and feasibility of HSCT using TCRαβ+/CD19+ depleted hematopoietic stem cells to treat non-malignant hematologic diseases. This will be assessed by evaluating the incidence of graft failure, grade III-IV acute GVHD and chronic GVHD and TRM. Secondary objectives include the evaluation of immune reconstitution and incidence of post-transplant infections, adverse events, serious adverse events, overall and disease-free survival and the efficiency of graft processing by the CliniMACS System.

ELIGIBILITY:
Inclusion Criteria:

* No Human leukocyte antigen (HLA) identical sibling available AND
* NO HLA matched unrelated donor available OR urgent need of HSCT precludes time necessary to search for suitable HLA matched unrelated donor AND
* Haploidentical donor OR closely matched unrelated donor available and willing to undergo mobilization and apheresis
* If subject has genetically confirmed inherited bone marrow failure, related donor must be evaluated for this disorder and testing must be negative.
* If subject has sickle cell disease, donor may have only sickle cell trait
* Patient must be diagnosed with one of the following diseases or disorders:

Hemoglobinopathies

* Sickle Cell Disease for patients ≤ 21 years of age for whom hydroxyurea has been trialed for at least six months, and failed
* Thalassemia Major for patients ≤ 21 years of age

Acquired Bone Marrow Failure Syndromes

* Paroxysmal Nocturnal Hemoglobinuria with bone marrow failure
* Myelodysplastic Syndromes (lower risk)

Inherited Bone Marrow Failure Syndromes

* Fanconi Anemia
* Diamond Blackfan Anemia
* Dyskeratosis Congenita and related telomere disorders
* Congenital Thrombocytopenia Syndromes
* Severe Congenital Neutropenia
* Shwachman-Diamond Syndrome
* Age ≤ 40 years (except patients with hemoglobinopathies)
* Life Expectancy ≥ 3 months
* Karnofsky (patients > 16 years)/Lansky (patients ≤ 16 years) index ≥ 60
* Organ Function Requirements

Renal Function

* Creatinine clearance or radioisotope Glomerular Filtration Rate (GFR) greater than or equal to 60 ml/min/1.73m^2

Liver Function

* Total bilirubin < 3 mg/dL
* Alanine aminotransferase (ALT)/ Serum glutamic-pyruvic transaminase; synonymous with ALT (SCPT) ≤ 3 x Upper Limit of Normal(ULN) for age

Cardiac Function

* Ejection fraction of > 40% by Multiple gated acquisition scan (MUGA) or echocardiogram

Pulmonary Function

* No evidence of dyspnea at rest
* No supplemental oxygen requirement
* If measured, carbon monoxide diffusion capacity (DLCO) > 50%
* Willing to use effective birth control method if patient is of reproductive potential
* Informed consent obtained (patient or legal representative)

Exclusion Criteria:

* Pregnant
* HIV infection
* Uncontrolled, serious active infection at screening
* Significant serious intercurrent illnesses
* Enrollment in any other treatment study that would interfere with the endpoints of this study according to judgement of Principal Investigator(or PI designee).

Ages: 3 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade III-IV acute graft-versus-host disease (GVHD) | 100 days post transplantation
  Acute GVHD will be assessed and graded according to the Keystone Consensus Criteria for staging and grading of acute graft-versus-host disease.
Incidence of extensive chronic GVHD | up to 2 years
  Chronic GVHD will be assessed according to the current CIBMTR (Center for International Blood and Marrow Transplant Research) manual reflecting a grading system published by Sullivan KM (Sullivan 1981).
Incidence of graft failure | up to 2 years after graft
  Graft failure - defined as failure to achieve ANC > 500 /µL at Day +28 or initial neutrophil engraftment followed by a decline in ANC < 500 /µL that is unresponsive to growth factor therapy (secondary graft failure).
Incidence of Treatment related mortality(TRM) | Day +100 post-HSCT
  TRM - defined as death from any cause other than disease progression.

SECONDARY OUTCOMES:
Time to neutrophil engraftment | up to 28 days following HSCT
  The time to neutrophil engraftment is defined as the post-transplant day that is the first of 3 consecutive days with an absolute neutrophil count (ANC) of >500/µL as assessed by CBC.
Time to platelet engraftment | up to 28 days following HSCT
  The time to platelet engraftment is defined as the post-transplant day that is the first of 3 consecutive days with a platelet count ≥ 20,000/µL as assessed by complete blood count(CBC), without platelet support (transfusion) for 7 days.
Percentage donor chimerism using Short tandem repeat (STR) | up to 12 months following HSCT
  Short tandem repeat (STR) analysis will provide the percentage donor chimerism at specific time points post-transplant.
Kinetics of lymphocyte reconstitution via immunophenotyping using flow cytometry | up to 12 months following HSCT
  Lymphocyte reconstitution will be assessed at specific time points post-HSCT, expressed as the percentage of white blood cells comprised of T, B and NK cell subsets.
CliniMACS system efficiency: Percentage of viable CD34+ cells recovered after the TCRαβ+ and CD19+ depletion procedure | up to 12 months following HSCT
CliniMACS system efficiency: log depletion value for CD19+ cells after the TCRαβ+ and CD19+ depletion procedure | Day 0
CliniMACS system efficiency: log depletion value of TCRαβ+ cells after the TCRαβ+ and CD19+ depletion procedure | Day 0
CliniMACS system efficiency: number of viable blood cell subsets after the TCRαβ+ and CD19+ depletion procedure | Day 0
  Number of viable CD34+ blood stem cells, CD20+ B cells, CD3-CD56+ NK cells, TCRαβ+ T cells, and TCRγδ+ T cells in the HSC graft after the TCRαβ+ and CD19+ depletion procedure
Correlation between GVHD incidence and donor killer-cell immunoglobulin-like receptor (KIR) haplotype content | up to 2 years
Correlation between GVHD incidence and killer-cell immunoglobulin-like receptor (KIR)/KIR-ligand mismatch between donor and recipient. | up to 2 years
Event free survival | up to 1 years
  An event is defined as death, graft failure or stable mixed chimerism with disease recurrence.
Overall survival (OS) | up to 2 years
Incidence of symptomatic bacterial/fungal and viral reactivation requiring therapy | up to 1 year
  The incidence of infections (symptomatic bacterial/fungal and viral reactivation requiring therapy) will be used as an additional safety measure
Number of participants with adverse events related to infusion of the HSC graft | Day 0
Incidence of serious adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Capitini, MD, Principal Investigator — University of Wisconsin, Madison; Jacques Galipeau, MD, Study Director — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No